CLINICAL TRIAL: NCT01823601
Title: A Cognitive-Behavioral Program Of Emotional Management and Feeling Of Psychological Well-Being
Brief Title: Behavioral Management and Psychological Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Estudos em Medicina Comportamental (Other)
Responsible Party: Principal Investigator, Prof.Dr.José Roberto Leite, Director, Centro de Estudos em Medicina Comportamental
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: UMC-04201301
Record Dates: First submitted 2013-03-30; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Psychological Well Being; Behavioral Management
Keywords: Well-Being; Life Management Program; Breathing; Meditation; Cognitive-Behavioral Training
MeSH Terms: conditions — Psychological Well-Being; Respiratory Aspiration | interventions — Health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seminars in Health (Active Comparator): This group of volunteers will attend to seminars in health. Each seminar will last about 120 minutes, a similar period of time used for training experimental group.
  Interventions: Behavioral: Seminars in Health
- Behavioral Management Program (Experimental): "Behavioral Management Program" consists in to teach to the volunteers procedures which involve autogenic muscle relaxation, progressive self-focus meditation and cognitive-behavioral training to change thoughts, beliefs and behavior in order to control emotions. This program will consist in 10 weekly sessions of about 120 minutes each.
  Interventions: Behavioral: Behavioral Management Program

INTERVENTIONS:
Behavioral: Behavioral Management Program — Consists in 10 Sessions of 120 minutes of duration, to train diaphragmatic breathing; autogenic training of muscle relaxation; progressive self-focus meditation and cognitive-behavioral training.
  Other Names: Life Management Program
  Arms: Behavioral Management Program
Behavioral: Seminars in Health — Volunteers that participate in 10 weekly sessions of seminars in health
  Arms: Seminars in Health

SUMMARY:
The aim of present study is to evaluate whether a program of behavioral and cognitive procedures for emotional control, and assertive training, produces well-being and improvement in quality of life of healthy volunteers.

DETAILED DESCRIPTION:
Healthy volunteers,not presenting neurologic or psychiatric disorders, 18 years or older,both genders, were selected, after a medical examination, to participate in the study. In a randomized controlled trial, the volunteers were submitted to sessions of muscle relaxation (autogenic method), progressive self-focus meditation, and cognitive-behavioral training in self-control of negatives feelings. They were also trained to determine goals and to determine each step to reach them (plan of action).The volunteers have to apply this strategy to control emotional behavior and improve interpersonal relationship. Anxiety and depression scores will be determined using the Beck self evaluation scales (BDI and BAI); quality of life will be determined using WHO-QOL inventory and the Ryff Scale will be used to measure Psychological Well-Being.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people, without neurological or psychiatry disorders, according to the results of a medical examination
* 18 years or older
* high school degree

Exclusion Criteria:

* Severe neurological or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Depression and Anxiety scores in Beck Depression Inventory and Beck Anxiety Inventory | Up to 3 month

SECONDARY OUTCOMES:
Evaluation of Well-Being scores in 6 factors of Psychological Well-Being in Ryff scale | Up to 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil